CLINICAL TRIAL: NCT04974944
Title: An Open-label, Phase 2 Randomized Trial of Camrelizumab (SHR1210) Plus Apatinib Versus Paclitaxel and Cisplatin/Carboplatin Plus Bevacizumab as a First-line Therapy in Patients With Stage IVB, Recurrent, or Persistent Cervical Cancer
Brief Title: First-line Treatment With Camrelizumab + Apatinib Versus Chemotherapy + Bevacizumab in Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-145-01
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Stage IVB Cervical Cancer; Recurrent Cervical Cancer; Persistent Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; apatinib; Paclitaxel; Cisplatin; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab + Apatinib (Experimental): On Day 1 and Day 15 of each 28-day cycle, participants receive an intravenous (IV) infusion of camrelizumab 200 mg Plus an oral apatinib 250 mg once daily. Apatinib will be administered 250 mg once every other day when completing twice tumor assessement. All treatments are administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Camrelizumab; Drug: Apatinib
- Paclitaxel + Cisplatin/Carboplatin + Bevacizumab (Active Comparator): On Day 1 of each 21-day cycle, participants receive an intravenous (IV) infusion of paclitaxel 175 mg/m^2 PLUS cisplatin 50 mg/m^2 WITH bevacizumab 15 mg/kg OR paclitaxel 175 mg/m^2 PLUS carboplatin Area Under the Curve (AUC) 5, WITH bevacizumab 15 mg/kg). All treatments are administered until disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Camrelizumab — IV injection
  Other Names: SHR1210
  Arms: Camrelizumab + Apatinib
Drug: Apatinib — Oral
  Arms: Camrelizumab + Apatinib
Drug: Paclitaxel — IV injection
  Arms: Paclitaxel + Cisplatin/Carboplatin + Bevacizumab
Drug: Cisplatin — IV infusion
  Arms: Paclitaxel + Cisplatin/Carboplatin + Bevacizumab
Drug: Carboplatin — IV infusion
  Arms: Paclitaxel + Cisplatin/Carboplatin + Bevacizumab
Drug: Bevacizumab — IV infusion
  Arms: Paclitaxel + Cisplatin/Carboplatin + Bevacizumab

SUMMARY:
Cervical cancer is the second-most common cancer in the world and is a leading cause of cancer death among women in developing countries. Cisplatin-based chemotherapy +/- bevacizumab have been recommended as the first-line treatment for patients who present with metastatic (e.g. stage IVB), persistent, or recurrent cervical cancer. However, patients in this setting are rarely curable. The immune checkpoint inhibitor (ICI) therapy, including cytotoxic T-lymphocyte antigen 4 (CTLA-4), programmed death-1 (PD-1), and programmed death-ligand 1 (PD-L1) inhibitors, has revolutionized the treatment of several cancers. The investigator previously reported the promising antitumor efficacy of camrelizumab (PD-1 inhibitor) combined with apatinib (VEGFR2 inhibitor) as second-line, or later, therapy in patients with advanced cervical cancer. This randomized study is to assess the efficacy and safety of first-line treatment with camrelizumab plus apatinib compared to the efficacy and safety of paclitaxel and cisplatin/carboplatin plus bevacizumab in patients with stage IVB, recurrent, or persistent cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Age ≥ 18 years and ≤ 70 years
* Patients must have primary stage IVB, recurrent or persistent squamous cell carcinoma of the cervix which has not been treated with systemic chemotherapy and is not amenable to curative treatment with surgery and/or radiation therapy NOTE: Prior adjuvant therapy is NOT counted as a systemic chemotherapeutic regimen for management of recurrent, persistent or metastatic carcinoma of the cervix; adjuvant therapy includes cisplatin given concurrent with primary radiation therapy (CCRT) and adjuvant chemotherapy given following the completion of concurrent chemotherapy and radiation therapy
* Patients must have measurable disease per RECIST v1.1; measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded as ≥ 10 mm with computed tomography (CT) scan, magnetic resonance imaging (MRI); a lymph node must be ≥ 15 mm in short axis. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* Life expectancy exceeds 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has the ability to swallow pills
* Provide cervical cancer tissue (archival or fresh biopsy specimen) prior to randomization for PD-L1 immunohistochemistry (IHC) testing by central laboratory
* Has PD-L1 IHC CPS ≥ 1 by central laboratory testing
* Has adequate organ function
* Female participants must not be pregnant, not breastfeeding. Female participants of childbearing potential should be willing to use one acceptable contraception (i.e., oral contraceptives, contraceptive injections, contraceptive implants, spermicides, condoms, intrauterine devices [IUDs]) during the treatment period and for 180 days following the end

Exclusion Criteria:

* Has an active autoimmune disease that has required systemic treatment; replacement therapy is not considered a form of systemic treatment.
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis;
* Has pleural effusion and ascites that require punctured and drained. However, an exception includes patients with pleural effusion and ascites who have no symptoms.
* Has bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage. Ureteral stent placement must be performed in patients with unilateral hydronephrosis prior to enrollment.
* Patients with a prior invasive malignancy who have had any evidence of disease within the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Clinically significant cardiovascular diseases, including but not limited to congestive heart failure (New York heart association (NYHA) class > 2), unstable or severe angina, severe acute myocardial infarction, or cardiac arrhythmia requiring medical intervention within 6 months before enrollment.
* Prior or concurrent diagnosis of idiopathic pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, and active pneumonia detected by CT during the screening period.
* Hypertension that can not be well controlled through antihypertensive drugs (systolic pressure ≥ 140 mm Hg and/or diastolic pressure ≥ 90 mm Hg)
* Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
* Patients have coagulation abnormalities with a tendency to bleed or are receiving thrombolytic or anticoagulant therapy. Prophylactic use of aspirin (≤100mg/d), low-molecular-weight-heparin (≤40mg/d), and Rivaroxaban is permitted.
* Any hemorrhage or bleeding event ≥ CTCAE Grade 2 within 4 weeks prior to the first dose of study intervention;
* Arterial thrombus or phlebothrombosis within 6 months prior to randomization.
* Gastrointestinal fistula, bladder/ureteral fistula, or intestinal obstruction within 6 months prior to randomization
* Has radiation-induced enteritis within 12 months prior to randomization
* Has received anticancer treatment, including but not limited to radiotherapy, chemotherapy, and surgery within 4 weeks before the first dose of study intervention
* Any unresolved toxicities (i.e., ≤ Grade 1 or at baseline) from prior therapy, with exception of alopecia;
* Has an active infection requiring systemic therapy or baseline white blood cells >1.5 × 10 9 / L;
* Has known active hepatitis B disease (hepatitis B virus [HBV] DNA > 500 IU/ml 1000 copies/ml) or hepatitis C disease;
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody, apatinib, and bevacizumab.
* Has a known history of human immunodeficiency virus (HIV) infection;
* Pregnant or breastfeeding.
* According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 36 months
  PFS defined as the time from randomization to the first documented disease progression per RECIST v1.1, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
  ORR is defined as the percentage of participants in the analysis population who have a complete response or a partial response per RECIST 1.1.
Duration of Response (DOR) | up to 24 months
  DOR is defined as the time from first documented evidence of CR or PR until disease progression per RECIST 1.1 or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | up to 24 months
  DCR is defined as the percentage of patients who have CR, PR, and stable disease (SD).
Overall Survival (OS) | up to 48 months
  OS is defined as the time from the treatment to death due to any cause.
Number of Subjects with treatment-related adverse events (AEs) | up to 48 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
Patient-reported outcomes (PROs) | up to 48 months
  PROs assessed by the Functional Assessment of Cancer Therapy-Cervix (FACT-Cx) Trial Outcome Index (TOI).
  The Functional Assessment of Cancer Therapy-General (FACT-G) is a 27-item self-report quality of life (QOL) measure that includes 4 subscales (physical well-being, social well-being, functional well-being and emotional well-being). The Trial Outcome of Index of FACT-Cx (FACT-Cx TOI) consists of two subscales from the FACT-G: Physical Well Being (7 items) and Functional Well Being (7 items), plus the Cervix Cancer-specific subscale (15 items). The total score is ranged 0-116 for FACT-Cx TOI. A higher score indicates better HRQL.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Huang, MD, Principal Investigator — Sun Yat-sen University Cancer Centre
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided